CLINICAL TRIAL: NCT05291871
Title: Immunogenicity of Fractional Dose of the HPV Vaccines
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Anna Wald, Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014983
Record Dates: First submitted 2022-03-03; First posted 2022-03-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HPV Infection; HPV Vaccine
Keywords: HPV, vaccines
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IM Bivalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of bivalent HPV vaccine administered intramuscularly
  Interventions: Biological: HPV vaccine
- ID Bivalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of bivalent HPV vaccine administered subcutaneously
  Interventions: Biological: HPV vaccine
- IM Nonavalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of nonavalent HPV vaccine administered intramuscularly
  Interventions: Biological: HPV vaccine
- ID Nonavalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of nonavalent HPV vaccine administered subcutaneously
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — One-fifth dose bivalent HPV Vaccine or One-fifth dose nonavalent HPV Vaccine

SUMMARY:
This randomized phase IV trial compares intramuscular and intradermal fractional dose of bivalent HPV vaccine to fractional dose of nonavalent HPV vaccine among men and women aged 27-45 years in Seattle, Washington. Participants will have immune response assessed at baseline, 4 weeks, 6 months, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Age 27-45 years at enrollment
* Not intending to receive the HPV vaccine series for the duration of the study participation
* Willing and able to: provide written informed consent, undergo clinical evaluation, adhere to follow-up schedule

Exclusion Criteria:

* Prior immunization with HPV-vaccine (Cervarix, Gardasil-4, Gardasil-9)
* Currently pregnant or breastfeeding
* Immunedeficiency disease/condition or cancer that causes clinically significant immunosuppression
* Known HIV infection
* Chemotherapy (current or within 12 months) or currently taking a medication that causes clinically significant immunosuppression.
* Unstable medical condition (e.g., malignant hypertension, poorly controlled diabetes)
* Known allergy to vaccine components
* Prior history of HPV-associated cancer
* Any medical condition which, in the opinion of the investigator, may compromise the subject's ability to safely complete the study.

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV antibody detection after intradermal or intramuscular, fractional one-fifth dose HPV-2 or HPV-9 vaccine immunization | 12 months
  To describe the changes in vaccine-type HPV antibody detection measured by Luminex assay between baseline and 12 months after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Stankiewicz Karita, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No